CLINICAL TRIAL: NCT03851874
Title: A Comparative Study of the Effects of Roux en Y Gastric Bypass and Sleeve Gastrectomy on Postprandial Gut Hormone Responses, Glycemia and Lipid Profile, Weight Loss, and Indices of Cardiovascular Risk
Brief Title: Comparison of Gastric Bypass and Sleeve Gastrectomy in Metabolic and Cardiovascular Indices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bariatric study
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Morbid Obesity
Keywords: Bariatric surgery, gut peptides, weight loss, glycemia
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric bypass bariatric surgery (Active Comparator): Patients in this arm underwent Roux-en-Y gastric bypass bariatric surgery for the treatment of morbid obesity
  Interventions: Procedure: Bariatric surgery
- Sleeve gastrectomy bariatric surgery (Active Comparator): Patients in this arm underwent sleeve gastrectomy bariatric surgery for the treatment of morbid obesity
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery

SUMMARY:
Morbidly obese patients undergoing either Roux en Y gastric bypass or sleeve gastrectomy were examined preoperatively, 3, 6, and 12 months after surgery. On each occasion, anthropometric data were collected, resting metabolic rate was measured, and the patients underwent a panel of cardiovascular examinations (heart rate variability, baroreflex sensitivity, heart ultrasound). Following that, they consumed a test meal and completed visual analog scales for the subjective assessment of hunger and fullness every 30 minutes for 3 hours. At the same time points, blood samples were collected for the consequent measurement of glucose, insulin, lipids, and gastrointestinal hormones.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 kg/m2
* Age between 18 and 65 years
* Proven failure to lose weight through non-surgical interventions

Exclusion Criteria:

* Serious and life threatening comorbidities (renal, cardiac, liver failure, or malignancy)
* Patients' inability to adhere to postsurgical instructions
* Alcohol or other substance abuse
* Concurrent psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in postprandial ghrelin responses | 3, 6, and 12 months
  Change in the cumulative postprandial response for ghrelin
Change in postprandial GLP-1 responses | 3, 6, and 12 months
  Change in the cumulative postprandial response for GLP-1
Change in postprandial PYY responses | 3, 6, and 12 months
  Change in the cumulative postprandial response for PYY

SECONDARY OUTCOMES:
Change in weight | 3, 6, and 12 months
  Change in weight (percentage of weight lost through each procedure)
Change in postprandial glycemia | 3, 6, and 12 months
  Change in the cumulative postprandial response for glucose
Change in postprandial insulinemia | 3, 6, and 12 months
  Change in the cumulative postprandial response for insulin
Change in postprandial triglyceridemia | 3, 6, and 12 months
  Change in the cumulative postprandial response for triglycerides

OTHER OUTCOMES:
Change in baroreflex sensitivity | 3, 6, and 12 months
  Changes in baroreflex sensitivity
Change in heart rate variability | 3, 6, and 12 months
  Changes in heart rate variability
Change in aortic distensibility | 3, 6, and 12 months
  Changes in aortic distensibility
Change in Tei index | 3, 6, and 12 months
  Changes in echocardiographic Tei index

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Kokkinos, MD, PhD, Principal Investigator — First Department of Propaedeutic Medicine, NKUA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holst JJ, Madsbad S. Mechanisms of surgical control of type 2 diabetes: GLP-1 is key factor. Surg Obes Relat Dis. 2016 Jul;12(6):1236-42. doi: 10.1016/j.soard.2016.02.033. Epub 2016 Mar 3. PMID 27313194
- [Background] Korner J, Bessler M, Inabnet W, Taveras C, Holst JJ. Exaggerated glucagon-like peptide-1 and blunted glucose-dependent insulinotropic peptide secretion are associated with Roux-en-Y gastric bypass but not adjustable gastric banding. Surg Obes Relat Dis. 2007 Nov-Dec;3(6):597-601. doi: 10.1016/j.soard.2007.08.004. Epub 2007 Oct 23. PMID 17936091
- [Background] Dimitriadis GK, Randeva MS, Miras AD. Potential Hormone Mechanisms of Bariatric Surgery. Curr Obes Rep. 2017 Sep;6(3):253-265. doi: 10.1007/s13679-017-0276-5. PMID 28780756
- [Background] Laferrere B, Swerdlow N, Bawa B, Arias S, Bose M, Olivan B, Teixeira J, McGinty J, Rother KI. Rise of oxyntomodulin in response to oral glucose after gastric bypass surgery in patients with type 2 diabetes. J Clin Endocrinol Metab. 2010 Aug;95(8):4072-6. doi: 10.1210/jc.2009-2767. Epub 2010 May 25. PMID 20501690
- [Background] Yousseif A, Emmanuel J, Karra E, Millet Q, Elkalaawy M, Jenkinson AD, Hashemi M, Adamo M, Finer N, Fiennes AG, Withers DJ, Batterham RL. Differential effects of laparoscopic sleeve gastrectomy and laparoscopic gastric bypass on appetite, circulating acyl-ghrelin, peptide YY3-36 and active GLP-1 levels in non-diabetic humans. Obes Surg. 2014 Feb;24(2):241-52. doi: 10.1007/s11695-013-1066-0. PMID 23996294
- [Background] Farey JE, Preda TC, Fisher OM, Levert-Mignon AJ, Stewart RL, Karsten E, Herbert BR, Swarbrick MM, Lord RV. Effect of Laparoscopic Sleeve Gastrectomy on Fasting Gastrointestinal, Pancreatic, and Adipose-Derived Hormones and on Non-Esterified Fatty Acids. Obes Surg. 2017 Feb;27(2):399-407. doi: 10.1007/s11695-016-2302-1. PMID 27465935
- [Derived] Angelidi AM, Kokkinos A, Sanoudou D, Connelly MA, Alexandrou A, Mingrone G, Mantzoros CS. Early metabolomic, lipid and lipoprotein changes in response to medical and surgical therapeutic approaches to obesity. Metabolism. 2023 Jan;138:155346. doi: 10.1016/j.metabol.2022.155346. Epub 2022 Nov 12. PMID 36375643